CLINICAL TRIAL: NCT06076564
Title: Leveraging Psychological Autopsies to Accelerate Research Into Stimulant Overdose
Brief Title: Leveraging Psychological Autopsies to Accelerate Research Into Stimulant Overdose Mortality
Acronym: LASSO
Status: Completed | Type: Observational
Sponsor: San Francisco Department of Public Health (Other Government)
Responsible Party: Principal Investigator, Phillip Coffin, MD, MIA, Director, Center on Substance Use and Health, San Francisco Department of Public Health
Other Study IDs: R01CE003364 (NIH)
Record Dates: First submitted 2023-09-22; First posted 2023-10-11 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Stimulant Overdose; Overdose Accidental; Overdose Cocaine; Overdose Methamphetamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Informants: Informants are individuals who knew someone who had a fatal stimulant overdose. Once a decedent is selected, their records will be reviewed to familiarize the interviewer with the situation of their death. Informants will be identified using contacts that the OCME used during their investigation, death records from the state, or emergency contacts from medical records, followed by recommendations from any of those contacts.
- Living Persons who use Stimulants: To identify resilience factors and risk reduction strategies among living persons who use stimulants, study staff will conduct interviews with up to 60 adults who use either cocaine or methamphetamine.

SUMMARY:
In the LASSO study, the investigators will identify 100 stimulant overdose decedents (divided among stimulant-only, and stimulant with fentanyl), conduct informant interviews (including scales and qualitative data), and gather data from the postmortem investigation (e.g., vital records, toxicology, autopsy, case narrative, death scene photographs) and medical record abstraction. Subsequently, study staff will conduct qualitative interviews with 40-60 living people who use stimulants (aiming for half methamphetamine, half cocaine) to explore elements of resilience and risk reduction strategies. This study aims to contribute to the eventual design of interventions to reduce stimulant overdose mortality.

DETAILED DESCRIPTION:
Death from acute stimulant toxicity ("overdose") is rapidly rising across the United States. While there are decades of research and program development undergirding opioid overdose prevention, there is minimal understanding of the nature of stimulant overdose mortality. Psychological autopsies have been shown to be immensely valuable in understanding opioid overdose deaths, identifying many of the key elements of overdose that still drive overdose prevention efforts today, and the investigators propose to leverage that mechanism to accelerate our understanding of and response to stimulant overdose mortality, as well as the role of fentanyl in fatal stimulant overdose.

The investigators will identify 100 stimulant overdose decedents (divided among stimulant-only, and stimulant with fentanyl), conduct informant interviews (including scales and qualitative data), and gather data from the postmortem investigation (e.g., vital records, toxicology, autopsy, case narrative, death scene photographs) and medical record abstraction. Subsequently, the study team will conduct qualitative interviews with 40-60 living people who use stimulants (aiming for half methamphetamine, half cocaine) to explore elements of resilience and risk reduction strategies. This study aims to contribute to the eventual design of interventions to reduce stimulant overdose mortality.

ELIGIBILITY:
Inclusion:

All informants must be at least 18 years of age and have knowledge of the decedent and that the decedent used substances.

If the contact has knowledge of the decedent's earlier life (e.g., family or long-term friend), the inclusion criteria are that they

1. are aware the decedent used substances in the past year prior the to date of death AND
2. have been in contact with the decedent in the past year prior to the date of death by phone, email, or in person

OR

If the contact has recent knowledge of the decedent (e.g., partners, friends, neighbors, or service providers), the inclusion criteria are that they

1. are aware the decedent used substances in the past 30 days prior to the date of death and
2. have been in contact with the decedent in person in the past year prior to the date of death.

Living persons who use stimulants:

1. ≥18 years of age,
2. Used cocaine or methamphetamine for ≥5 years,
3. Used cocaine or methamphetamine for ≥10 out of the past 30 days, AND
4. Matched to a decedent on age, race/ethnicity, gender, and neighborhood distribution of decedents of the methamphetamine/no opioid and cocaine/no opioid decedents.

Exclusion:

Informants:

No exclusion criteria.

Living persons who use stimulants:

1. Used both cocaine and methamphetamine ≥5 of past 30 days,
2. Intentionally use illicit opioids, OR
3. Unable to communicate in English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All informants must be at least 18 years of age and have knowledge of the decedent and that the decedent used substances. Living persons who use stimulants must be at least 18 years of age and use cocaine or methamphetamine.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Clinical antecedents to stimulant overdose. | One year prior to the date of death.
  The investigators will use medical records and mortality data, as well as qualitative and quantitative interview data with close contacts, to identify medical, psychological, and substance use antecedents to stimulant overdose death.
Antecedent patterns between stimulant overdose deaths with and without fentanyl. | One year prior to the date of death.
  The investigators will compare stimulant (without fentanyl) deaths to stimulant with fentanyl deaths to identify key differences, such as in substance use, suicidality, cardiac and other medical or psychiatric events, between the two groups.
Resilience factors and risk reduction strategies among living persons who use stimulants. | One year prior to the interview date.
  The investigators will use quantitative and qualitative data obtained from interviews with people who use stimulants to identify resilience and risk reduction strategies that reduce the risk for fatal stimulant overdose.

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Department of Public Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No